CLINICAL TRIAL: NCT03221842
Title: A Double-blind, Randomized-withdrawal, Placebo-controlled Study to Evaluate the Efficacy and Safety of Human Plasma-derived C1-esterase Inhibitor as add-on to Standard of Care for the Treatment of Refractory Antibody Mediated Rejection in Adult Renal Transplant Recipients
Brief Title: Efficacy and Safety of Human Plasma-derived C1-esterase Inhibitor as add-on to Standard of Care for the Treatment of Refractory Antibody Mediated Rejection (AMR) in Adult Renal Transplant Recipients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated early due to futility of enrolment and not for safety reasons.
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSL842_3001; 2017-000348-17 (EudraCT Number)
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Results first posted 2022-01-18 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Antibody-mediated Rejection
Keywords: Antibody-mediated kidney transplant rejection; Renal
MeSH Terms: interventions — Complement C1 Inhibitor Protein

STUDY DESIGN:
Intervention Model Description: Randomized-withdrawal
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- C1-INH (Experimental): C1-esterase inhibitor
  Interventions: Drug: C1-esterase inhibitor
- Placebo (Placebo Comparator): Excipients of C1-INH plus albumin
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: C1-esterase inhibitor — C1-esterase inhibitor is a human plasma-derived lyophilised powder for reconstitution
  Other Names: C1-INH
  Arms: C1-INH
Drug: Placebo — Excipients of C1-INH plus albumin
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized-withdrawal, placebo-controlled study in kidney transplant patients with AMR to evaluate the efficacy and safety of human plasma-derived C1-esterase inhibitor as add-on to standard of care (IVIG).

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age;
* Evidence of at least one donor-specific antibody (DSA);
* Recipient of a kidney transplant;
* Achieved a steady-state, post-transplant eGFR ≥ 40 mL/min/1.73 m2 within 60 days of post-transplant OR a 50% increase in urine output with a 50% decrease in serum creatinine over the first 7 days post-transplant in subjects with slow or delayed graft function;
* Acute AMR.

Exclusion Criteria:

* Recipient of an en bloc kidney transplant;
* Current active hepatitis C virus (HCV) infection;
* Active bacterial or fungal infection;
* Ongoing dialysis >2 weeks;
* Known congenital bleeding or coagulopathy disorder;
* Current cancer or a history of cancer;
* Female subjects who are pregnant or breast feeding;
* Male or female subjects who are unwilling to use contraception or who are not surgically sterile.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Program Director, Study Director — CSL Behring
Locations (26):
- United States (13):
  - University of Alabama Hospital (at Birmingham), Birmingham, Alabama
  - Mayo Clinic Arizona, Phoenix, Arizona
  - California Pacific, San Francisco, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - University of Illinois Chicago, Chicago, Illinois
  - Brigham & Women's, Boston, Massachusetts
  - Mayo Clinic (Rochester), Rochester, Minnesota
  - St. Barnabas Medical Center, Livingston, New Jersey
  - NYU, New York, New York
  - Columbia University, New York, New York
  - Vanderbilt University, Nashville, Tennessee
  - Houston Methodist, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin
- Universitair Ziekenhuis Gasthuisberg, Leuven, Belgium
- France (7):
  - CHU de Bordeaux. Hôpital Pellegrin, Bordeaux
  - CHU de Grenoble - Hôpital Michalon, Grenoble
  - Centre Regional Hospitalier Universitaire de Lille, Lille
  - Hospital Edouard Herriot Lyon, Lyon
  - Hopital saint Louis Paris, Paris
  - Necker Hospital, Paris
  - CHU Rangueil, Toulouse
- Charite Berline, Berlin, Germany
- Leiden University Medical Center, Leiden, Netherlands
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
- Guy's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Viklicky O, Slatinska J, Novotny M, Hruba P. Developments in immunosuppression. Curr Opin Organ Transplant. 2021 Feb 1;26(1):91-96. doi: 10.1097/MOT.0000000000000844. PMID 33332922

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only 13 participants that completed Period 1 were eligible to continue to Period 2. Eligibility based on the amendment in place at the time the subject completed Period 1.
Groups:
- C1-INH: C1-esterase inhibitor (CSL842)
  C1-esterase inhibitor: C1-esterase inhibitor is a human plasma-derived lyophilised powder for reconstitution administered at a dose of 60 IU/kg
Period: Period 1 (Open-label)
Arm/Group | C1-INH | Placebo
Started | 63 | 0
Completed | 53 | 0
Not Completed | 10 | 0
Not completed — Adverse Event | 4 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Terminated by sponsor | 1 | 0
Not completed — Other | 2 | 0
Period: Period 2 (Randomized, Blinded)
Arm/Group | C1-INH | Placebo
Started | 7 | 6
Completed | 6 | 5
Not Completed | 1 | 1
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Arm/Group | C1-INH
Number analyzed (Participants) | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (13.83)
Age, Customized [Number; unit: participants]
  >=18 and <65 years | 57
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 52
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 39
  More than one race | 1
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Loss-of-response During Treatment Period 2 (TP2)
Description: Loss of response is defined as 1 of the following, whichever occurs first:
  * Decline in Estimated Glomerular Filtration Rate (eGFR), or
  * Allograft failure, or
  * Subject death by any cause.
Time Frame: Up to 38 weeks
Population: Modified Intent-to-Treat Analysis Set (mITT) - All subjects randomized under the original protocol and under all protocol amendments were included in this population except the subjects randomized prior to Amendment 3 who did not satisfy the responder criteria updated in Amendment 3.
Measure: Number; unit: percentage of participants
Arm/Group | C1-INH | Placebo
Number analyzed (Participants) | 6 | 5
percentage of participants | 33.3 | 40.0

2. Secondary Outcome: Number of Participants With All-cause Allograft Failure During TP2
Description: Allograft failure is defined as 1 of the following:
  * Allograft nephrectomy, institution of permanent dialysis, or return to the transplant waitlist for renal transplant, whichever occurs first, OR
  * Subject death by any cause
Time Frame: Up to 38 weeks
Population: mITT
Measure: Number; unit: number of participants
Arm/Group | C1-INH | Placebo
Number analyzed (Participants) | 6 | 5
number of participants | 0 | 1

3. Secondary Outcome: Percent of Participants With All-cause Allograft Failure During TP2
Time Frame: Up to 38 weeks
Population: mITT
Measure: Number; unit: percentage of participants
Arm/Group | C1-INH | Placebo
Number analyzed (Participants) | 6 | 5
percentage of participants | 0 | 20

4. Secondary Outcome: Absolute Change From Baseline in Estimated Glomerular Filtration Rate at End of Treatment Period 1 (TP1)
Time Frame: Baseline and 13 weeks
Population: The Run-in Safety (RiS) analysis set comprised all subjects who received at least 1 dose of C1-INH during TP1.
Measure: Median (Full Range); unit: mL/min/1.73m^2
Arm/Group | C1-INH
Number analyzed (Participants) | 63
mL/min/1.73m^2 | -0.75 [-17.0 to 7.5]

5. Secondary Outcome: Absolute Change From Baseline in Estimated Glomerular Filtration Rate at End of TP2
Time Frame: Baseline and 38 weeks
Population: mITT
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | C1-INH | Placebo
Number analyzed (Participants) | 6 | 4
mL/min/1.73m^2 | 7.75 (8.454) | 15.25 (10.444)

6. Secondary Outcome: The Rate of Change of eGFR During TP2 as Defined by the Slope of the Mean Regression of eGFR Over Time at End of TP2
Description: The Sponsor terminated the study due to futility of enrolment. Because of the study termination, limited efficacy results are presented in this report.
Time Frame: Up to 38 weeks
Population: The Sponsor terminated the study due to futility of enrolment. Because of the study termination, limited efficacy results are presented in this report. Due to study termination, data was not collected for this endpoint.
Arm/Group | C1-INH | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Time to All-cause Allograft Failure Through the Follow up Period
Description: as for outcome 6
Time Frame: Up to approximately 208 weeks
Population: as for outcome 6
Arm/Group | C1-INH | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Responders at the End-of-TP1
Description: Responders were defined as subjects whose End-of-TP1 eGFR was ≥ 90% of baseline eGFR and ≥ 20 mL/min/1.73 m2.
Time Frame: Up to 13 weeks
Population: RiS
Measure: Number; unit: participants
Arm/Group | C1-INH
Number analyzed (Participants) | 63
participants | 33

9. Secondary Outcome: Percent of Responders at the End-of-TP1
Description: Responders were defined as subjects whose End-of-TP1 eGFR was ≥ 90% of baseline eGFR and ≥ 20 mL/min/1.73 m2.
Time Frame: Up to 13 weeks
Population: RiS
Measure: Number; unit: percentage of responders
Arm/Group | C1-INH
Number analyzed (Participants) | 63
percentage of responders | 52.4

10. Secondary Outcome: Proportion of Subjects Surviving Through the Follow-up Period
Description: as for outcome 6
Time Frame: Up to approximately 208 weeks
Population: as for outcome 6
Arm/Group | C1-INH | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Percent of Participants With Any Adverse Event (AE) Assessed as Related to Investigational Product
Time Frame: Up to approximately 42 weeks after the time of first investigational product administration
Population: RiS and RWS [The Randomized Withdrawal Safety (RWS) analysis set included all subjects in the ITT analysis set who received at least 1 dose of the investigational product after randomization during TP2]
Measure: Number; unit: percentage of participants
Groups:
- C1-INH (Period 1); C1-INH (Period 2): C1-esterase inhibitor (CSL842)
  C1-esterase inhibitor: C1-esterase inhibitor is a human plasma-derived lyophilised powder for reconstitution administered at a dose of 60 IU/kg
Arm/Group | C1-INH (Period 1) | C1-INH (Period 2) | Placebo
Number analyzed (Participants) | 63 | 7 | 6
percentage of participants | 20.6 | 0 | 16.7

12. Secondary Outcome: Mean Pre-dose C1-esterase Inhibitor Functional Activity
Description: C1-esterase Inhibitor may play a role in the prevention of antibody-mediated rejection (AMR) following kidney transplant. Low levels of C1 esterase inhibitor concentration and its functional activity may lead to AMR. Patients with AMR may go on to lose their kidney transplant and have other associated health risks. Levels of C1-esterase inhibitor functional activity in plasma is described as a percent.
Time Frame: Up to 13 weeks
Population: The pharmacokinetic analysis set (PK) comprised all subjects who consented to provide rich PK sampling, who received ≥ 1 dose of C1-INH, and who had ≥ 1 measurable level of C1-INH functional activity. (some participants had missing data) or C1-INH antigen concentration.
Measure: Mean (Standard Deviation); unit: percent functional activity
Arm/Group | C1-INH
Number analyzed (Participants) | 20
percent functional activity
  week 2: number analyzed (Participants) | 14
  week 2 | 168.86 (64.059)
  week 11: number analyzed (Participants) | 13
  week 11 | 179.32 (58.551)

13. Secondary Outcome: Area Under the Plasma Concentration Time Curve (AUC0-t) for C1-INH Functional Activity
Description: C1-esterase Inhibitor may play a role in the prevention of antibody-mediated rejection (AMR) following kidney transplant. Low levels of C1 esterase inhibitor concentration and its functional activity may lead to AMR. Patients with AMR may go on to lose their kidney transplant and have other associated health risks. Levels of C1-esterase inhibitor functional activity is described as a percent.
Time Frame: Up to 72 hours after post-dose on Day 10 and on Day 77 of Period 1
Population: PK (some participants had missing data)
Measure: Mean (Standard Deviation); unit: hours*percent functional activity
Arm/Group | C1-INH
Number analyzed (Participants) | 15
hours*percent functional activity
  Day 10: number analyzed (Participants) | 10
  Day 10 | 15229.84819 (4149.16754)
  Day 77: number analyzed (Participants) | 9
  Day 77 | 12742.20883 (4445.31881)

14. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) for C1-INH Functional Activity
Time Frame: Up to 72 hours after post-dose on Day 10 and on Day 77 of Period 1
Population: PK (some participants had missing data)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | C1-INH
Number analyzed (Participants) | 15
hours
  Day 10: number analyzed (Participants) | 14
  Day 10 | 9.9298 (16.3288)
  Day 77: number analyzed (Participants) | 10
  Day 77 | 37.9251 (22.8543)

ADVERSE EVENTS:
Time Frame: Up to 42 weeks per participant
Groups:
- Placebo (Period 2): Excipients of C1-INH plus albumin
  Placebo: Excipients of C1-INH plus albumin
Arm/Group | C1-INH (Period 1) | C1-INH (Period 2) | Placebo (Period 2)
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/7 | 1/6
Serious Adverse Events (participants affected / at risk) | 25/63 | 1/7 | 3/6
Other Adverse Events (participants affected / at risk) | 46/63 | 4/7 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | C1-INH (Period 1) (N=63) | C1-INH (Period 2) (N=7) | Placebo (Period 2) (N=6)
Blood creatine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Transplant rejection (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Unevaluable event (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Perinephric collection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pyelocaliectasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacterial pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urethritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound infection pseudomonas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | C1-INH (Period 1) (N=63) | C1-INH (Period 2) (N=7) | Placebo (Period 2) (N=6)
Hypertension (Vascular disorders) | 6 (7) | 1 (1) | 0 (0)
Refractory cytopenia with unilineage dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 4 (4) | 1 (1) | 0 (0)
Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 8 (9) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (4) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 5 (5) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 8 (9) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 5 (7) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (10) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 18 (32) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 11 (23) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (12) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 11 (13) | 0 (0) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 5 (5) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 0 (0) | 0 (0)
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Dermatitis papillaris capillitii (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Folate deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 5 (6) | 1 (1) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 3 (3) | 1 (2) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Trichomoniasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The Sponsor terminated the study due to futility of enrolment. Because of the study termination, there are limitations in interpreting analyses and efficacy results based on small numbers of subjects. No subject reached the 48-month follow-up endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/42/NCT03221842/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT03221842/SAP_001.pdf